CLINICAL TRIAL: NCT06628388
Title: Nurse-led Primary Healthcare Intervention Model in Women's Health Management in Hong Kong
Acronym: JCDATAZONEWH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); Haven of Hope Hospital (Other); Hong Kong Sheng Kung Hui Welfare Council Limited (Other); Aberdeen Kai-fong Welfare Association (Other)
Responsible Party: Principal Investigator, Prof. Sophia Siu-chee Chan, Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UW 24-501
Record Dates: First submitted 2024-09-27; First posted 2024-10-08 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Vasomotor Symptoms; Urinary Incontinence; Anxiety; Depression - Major Depressive Disorder; Osteoporosis; Breast Cancer; Hypertension; Cervical Cancers; Colorectal Cancer
Keywords: nurse-led; women health; risk-based; primary healthcare; 5As model; stepped-wedge; cluster RCT; health resource utilization; self-management; risk stratification; health screening
MeSH Terms: conditions — Urinary Incontinence; Anxiety Disorders; Osteoporosis; Breast Neoplasms; Hypertension; Uterine Cervical Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomized waitlist-controlled trial will be conducted. Stepped-wedge design is considered as a unidirectional crossover RCT. Current trial will consist of four consecutive phases with each lasting for four months. The three social service organizations will be the three clusters to be randomized. In the first phase, all participants in all three clusters will be allocated to the waitlist-control treatment. In the second phase, newly joined participants in cluster 1, randomly determined, will be exposed to the intervention condition, while the other two clusters remain in the waitlist-control. In the third phase, newly joined participants in cluster 1 and 2, will be allocated to the intervention condition, while cluster 3 remain receiving the waitlist-control condition. In the fourth phase, all newly recruited participants in the three clusters will be allocated to intervention condition.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal intervention (Active Comparator): Participants allocated to the control group condition will be given minimal intervention in standard practices at baseline and 3-month. It consist of general health education and advice, where the health information is open resources available for the public. No risk-stratified services nor active referral will be conducted by nurse until 6-month assessment is completed. After that, they will immediately receive intervention based on their 6-month assessment, and booster interventions at 7-month contact and 12-month follow-up.
  Interventions: Behavioral: Minimal Intervention
- Nurse-led Risk-based 5As Intervention Arm (Experimental): Participants allocated to the intervention condition will receive the nurse-led 5As model intervention at baseline, 1- and 3-month boosters, and 6- and 12-month follow-ups. The current model includes risk assessments and stratification, general health education booklet, consultations and active referrals based on personal risk stratification at baseline and 3-month booster, with additional booster session at 1-month, and follow-up sessions at 6- and 12-month from baseline. For participants with high risk of any target health conditions at baseline and 3-month booster, medical referral and service utilization (e.g., GPs/network doctors/specialist consultation at health centres/hospitals/clinics, screening, therapies, corresponding District Health Centre schemes, etc.) will be arranged at the visits. Such medical resource utilization among participants will be encouraged and motivated at 1-month booster session.
  Interventions: Behavioral: Nurse-Led Risk-Based 5As Primary Healthcare Model

INTERVENTIONS:
Behavioral: Nurse-Led Risk-Based 5As Primary Healthcare Model — The intervention is developed based on the 5As model (ask, advice, assess, assist, arrange). In this model, nurse will play the central role in delivering the service as a case manager. In Ask, all participants will be assessed on the demographics, health related status, and health risk stratification (i.e. 3-tier risk stratification). In Advice, all participants will be given the education booklet. Those assessed to be at low risks will receive general advice, while those at medium risk will receive condition-specific advice instead. High risk participants will be provided with referral suggestions. The assessment of medium or high risk participants willingness and any barriers in seeking changes will be conducted in Assess. In Assist, active referrals will be provided to high risk participants, with weekly advice messages provided to medium and high risk participants. In Arrange, all participants will receive their follow-ups.
  Arms: Nurse-led Risk-based 5As Intervention Arm
Behavioral: Minimal Intervention — Consisting general advice on women health with the education booklet. No risk-based services nor active referral will be offered during the waitlist control exposure. Participants will be switched to receive intervention from 6-month.
  Arms: Minimal intervention

SUMMARY:
The goal of this randomized clinical trial is to learn if a nurse-led primary healthcare intervention can help improve health management in women adults aged 45 to 64, and to develop an evidence-based primary healthcare model for women. The questions it aims to answer are:

if the intervention improves medical resource use, especially at 3-month from the beginning of intervention? if the intervention improves health confidence, self-management, and quality-of-life? if the intervention improves health conditions as reflected by risk levels?

Researchers will compare the intervention with the control group over time to see if there are better medical resource use, health confidence, self-management, and quality-of-life, and health conditions risk levels.

All participants will be asked to answer a set of questionnaires assessing their social demographics, health-related status, and risk levels of the targeted health conditions. All participants will receive an education booklet containing essential knowledge and available medical resources. Participants in the intervention group will receive nurse-led 5As (ask, advice, assess, assist, arrange) intervention which offers risk-specific health services. Participants will be followed at 3-, 6-, 12-month; with high risk participants will be followed additionally at 1-month after the beginning of intervention. Participants in the waitlist control group will be given general health advice as minimal intervention, followed-up at 3- and 6-month, provided with intervention of the same content with intervention group at 6-month, followed-up at 7-month and 12-month.

DETAILED DESCRIPTION:
Background:

Globally, the aging population is on the rise, leading to the phenomenon known as the "feminization of aging" (United Nations, 2017). In most regions, women outlive men and face an increased risk of severe illnesses and multiple health conditions, significantly impacting their quality of life (Chłoń-Domińczak et al., 2014). In Hong Kong, the Family Health Service of the Department of Health provides the Woman Health Services including health assessment, health education, and individual counseling at three Woman Health Centres (WHCs) to women aged at or below 64 years, and its coverage is very limited. Hence, there is a lack of evidence-based services in primary healthcare settings such as DHCs for identifying and stratifying health risks among women and effective interventions in promoting women's health, particularly for those older female adults.

Nurse-led intervention is an intervention where nurses play central roles and have autonomous rights in decision-making as well as authority in customizing patient care (Li et al., 2020). Despite the important role of nurses in primary health care, this is no innovative nurse-led intervention model targeting women's health in Hong Kong.

The '5As model', which was initially developed for smoking cessation based on changes to different stages within the healthcare intervention (Wang et al., 2019), consists of five main steps: identifying health status and behavior for each individual (Ask), advising and urging the behavioral changes (Advice), assessing the willingness and readiness to change (Assess), providing supports and referrals to individuals willing to change (Assist), and scheduling follow-ups to address barriers and discuss personal progress (Arrange). It has been found to be an effective and simple model for nurses to deliver healthcare promotion and education intervention in community (Kolac et al., 2023; Slev et al., 2020). Brief intervention model as such would be much more feasible in PHC settings (Saitz et al., 2010).

As women reach the middle stage of their life between the ages of 45 and 64, a significant number of them undergo hormonal changes linked to the transitions through menopause. These changes often lead to the emergence of novel health challenges (Nasreen et al., 2021). Apart from the commonly observed age-related risk of developing colorectal cancer, more prevalent conditions affecting women in this life phase are vasomotor symptoms (VMS), urinary incontinence (UI), depression and anxiety, osteoporosis, breast cancer, hypertension, and cervical cancer. Hence, based on the 5As model, a nurse-led risk-based primary healthcare intervention is proposed for women's health management in Hong Kong.

Study Design:

A stepped-wedge cluster randomized waitlist-controlled trial (SWT) will be conducted. The study period will consist of four consecutive phases with each lasting for four months. The three social service organizations will be the three clusters to be randomized. In the first phase, all participants in all three clusters will be allocated to the waitlist-control treatment. In the second phase, newly joined participants in cluster 1, randomly determined, will be exposed to the intervention condition, while the other two clusters remain in the waitlist-control. In the third phase, newly joined participants in cluster 1 and 2, will be allocated to the intervention condition, while cluster 3 remain receiving the waitlist-control condition. In the fourth phase, all newly recruited participants in the three clusters will be allocated to intervention condition. At 6-month follow-up, the waitlist-control participants will be given the same treatment as in intervention condition. A web-based portal system will be created for nurses to facilitate better case management and client coordination.

Procedures:

The NGO staff will receive two day training on clinical knowledge, health condition specific advice and appropriate community medical resources, behavioral modification skills, and study workflow. Booster training the study flow, risk assessment, and use of the web-based portal system will be provided during transition period. Service units of the three non-governmental organizations (NGOs) in the three districts (Aberdeen Kai Fong Association in Southern District (AKA), Haven of Hope Christian Services in Sai Kung District (HOHCS), and Hong Kong Sheng Kung Hui Welfare Council Limited in Wong Tai Sin District (SKHWC)) will screen and recruit appropriate participants for this trial. Recruitment ads will be posted onto offline (e.g., on-site posters) and online platforms (e.g., Facebook and Instagram). Women aged between 45 and 64 will be continuously recruited in the 4 recruitment phases. Participants would include but not limited to those who that are regular attendees (e.g., members) of the three social service organizations, and those in the general population who are seeking primary healthcare services through various offline/online recruitment approaches. Participants will undergo eligibility screening following registration. Eligible participants with consents will be enrolled in the current stepped-wedge waitlist-control randomized trial. For participants who do not meet the eligibility criteria for the current trial but express their willingness in receiving primary healthcare services, such rights will be protected and healthcare services/resources in need will be provided.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong female residents aged 45 to 64 years old; and
2. Able to read and communicate in Chinese (either Cantonese or Mandarin).

Exclusion Criteria:

1. Have a terminal illness (e.g., advanced cancer, dementia, pulmonary, neurological, motor-neuron, and advanced cardiovascular disease), or with a life expectancy of less than six months;
2. Diagnosed with psychiatric or psychological disorders (e.g., panic disorder, psychosis);
3. Currently taking medication(s) or receiving treatment(s) for psychiatric and psychological disorders;
4. Pregnant or in lactation period, or have plans for pregnancy within 1 year; or
5. Have moderate or severe cognitive impairment.

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1728 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Rate of medical resource utilization | 3-month from baseline
  Defined as completion of any referral (Women Health Centres or Maternal and Child Health Centres listed by the Depratment of Health, Kwong Wah Hospital Well Women Clinic, Tung Wah Group of Hospitals Well Women Clinic (North Point), Hong Kong Adventis Hospital Well Women Clinic, Women's Health Service by The Family Planning Association of Hong Kong, Canossa Hospital Health Check Centre, Primary Healthcare Directory Doctors, Hong Kong Breast Cancer Foundation Jockey Club Holistic Breast Health Project, Chronic-Disease Co-Care Pilot Scheme by Distric Health Centres, Colorectal Cancer Screenings (including Fecal Occult Blood Test, Sigmoidoscopy, or Colonoscopy), Jockey Club Holistic Support Project for Elderly Mental Wellness (JC JoyAge), or Integrated Community Centre for Mental Wellness) for consultation, prescriptions, screening, therapy, etc targeting health condition of concerns. A binary result with either "Yes" or "No" will be recorded.

SECONDARY OUTCOMES:
Rate of medical resource utilization | 1- , 6-, 7-, and 12-month after baseline.
  Defined as completion (with response 'Yes' or 'No') of any medical referral (to corresponding referral sites) for consultation, prescriptions, screening, therapy, etc targeting health condition of concerns. A binary result with either "Yes" or "No" will be recorded.
Characteristics of medical resource utilization | 1- , 6-, 7-, and 12-month after baseline.
  Defined as the detailed information on service goal (i.e. as preventive care or treatment), targeted health conditions, date and result of screenings, number of times of consultation or therapy session.
Score of self-reported Health Confidence Scale (HCS) | 1- , 3-, 6-, 7-, and 12-month after baseline.
  Self-reported health confidence will be measured using the Health Confidence Scale (HCS) consists of four items, each has four response options (score 3 as strongly agree, 2 as agree, 1 as neutral, 0 as disagree). Total score of the scale ranging from 0 to 12, higher score indicates better response. After transposing to a 0 to 100 scale, the score is categorized as very low (transposed score 0-39), low (transposed score 40-59), medium (transposed score 60-79), high (transposed score 80-100).
Score of self-reported Self-Management Assessment Scale (SMASc) | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The self-reported health management will be assessed using the Self-Management Assessment Scale (SMASc) consists of 10 items each with a 6-point Likert scale ranging from score 1 as strongly disagree to score 6 as totally agree. The 10 items were divided into five aspects, each aspect contains 2 items. Total score of each aspect ranging from 2 to 12, higher score indicates better response. Mean score of each aspect is categorized immediate need for self-management support (mean score 1-4), no acute need for self-management support (mean score 5-8), no need for self-management support (mean score 9-12).
Score in HK Chinese version of the EQ-5D-5L instrument (EQ-5D-5L HK) measuring quality of life | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The quality of life will be asse ssed using the HK Chinese version of the EQ-5D-5L instrument (EQ-5D-5L HK) consists of self-reported health on a 5-dimension descriptive system, each with 5 level of severity ranging from score 1 as no problem to score 5 as experiencing extreme problems. For the EQ-5D-5L HK, the overall response ranges from 11111 as full health, to 55555 as the worst health.
Score in EuroQol Visual Analogue Scale (EQ-VAS) measuring quality of life | 1- , 3-, 6-, 7-, and 12-month after baseline.
  As a generic health-related quality of life (HRQoL) measure, the EuroQol Visual Analogue Scale (EQ-VAS) will be used to assess patients global subjective well-being. For EQ-VAS, the overall score ranging from 0 as the worst health to 100 as the best health.
Risk level of vasomotor symptoms | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The vasomotor symptoms risk level will be assessed using the VMS 2Q scale consists of 2 items each with 5 response ranging from score 0 as none, score 1 as 1 to 5 days/2 weeks, score 2 as 6 to 8 days/2 weeks, score 3 as 9 to 13 days/2 weeks, to score 4 as everyday/2 weeks. The risk level is categorized as low risk (both items scored 0), medium (either item scored 1), high (either item scored 2 or more).
Types of urinary incontinence | 1- , 3-, 6-, 7-, and 12-month after baseline.
  Urinary incontinence types will be assessed using the 3 Incontinence Questionnaire consisting of 3 items in differentiating the types of urinary incontinence (i.e. stress only or stress predominant, urge only or urge predominant, other cause only or other cause predominant, mixed).
Risk level of urinary incontinence | 1- , 3-, 6-, 7-, and 12-month after baseline.
  Urinary incontinence severity will be assessed using the Incontinence Severity Index consisting of 2 items assessing the urinary incontinence frequency (ranging from score 0 as never; to score 4 as every day and/or night) and amount (ranging from score 0 as never; to score 4 as more). Total score equals to score of item 1 times item 2, ranging from 0 to 12. Total index score is defined as none (0), slight (1-2), moderate (3-6); severe (8-9); very severe (12). The risk level is categorized as low (scored 2 or lower), medium (scored 3-6), high (scored 8 or higher).
Risk level of depression | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The depression levels will be assessed using the Patient Health Questionnaire-9 consists of 9 items each with 4 responses ranging from score 0 as not at all to 3 as nearly every day. Total score ranges from 0 to 27, defined as mild (cutoff score of 5), moderate (cutoff score of 10), moderately severe (cutoff score of 15), severe (cutoff score of 20). The risk level is categorized as low (scored 4 or less), medium (scored 5-9), and high (scored 10 or more).
Risk level of anxiety | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The anxiety risk level will be assessed using the Generalized Anxiety Disorder 2-item consists of 2 items with responses ranging from score 0 as not at all to 3 as nearly every day. Total score ranges from 0 to 6, with a score greater or equal to 3 denotes a clinically significant anxiety. The risk level is categorized as low (scored 1 or less), medium (scored 2), and high (scored 3 or more).
Risk level of osteoporosis | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The risk level of osteoporosis will be assessed via the Chinese Osteoporosis Screening Algorithm (with response of score ≤ 0 or score greater than 0) together with the BeeTLE devices (with T-score ≥ -1, -1 to -2.5, or ≤ -2.5 for post-menopausal women; or Z-score < 0 or equal to or greater than -2.0 for pre-menopausal women). Risk levels are categorized as low (COSA≤ 0 and T-score ≥ -1.0 / Z-score greater than or equal to 0; or anyone with normal DXA scores as defined by the The Osteoporosis Society of Hong Kong https://oshk.org.hk/osteoporosis-risk-factor/ and NIH https://www.niams.nih.gov/health-topics/bone-mineral-density-tests-what-numbers-mean), medium (T-score -2.5 to -1.0, or those with COSA less or equal to 0 but BeeTle Z-score<0), and high (COSA greater than 0, or T-score ≤ -2.5; or anyone with osteoporosis DXA score).
Risk level of breast cancer | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The breast cancer risk level will be assessed using the assessment questionnaires and online calculation tools (www.cancer.gov.hk/bctool). For those who are suitable to for tool risk assessments, the risk percentage will be calculated as ≤25%, 26-50%, 51-75%, 76-99%, or greater than 99%. Risk levels are categorized as low (tool assessed risk ≤25%; or anyone with valid negative mammography results as defined by CEWG), medium (tool assessed risk 26%-75%), high (tool assessed risk ≥ 76%, or those unsuitable for the tool who meet the Hong Kong Cancer Expert Working Group high or moderate risk factors as described in https://www.chp.gov.hk/files/pdf/breast_cancer_professional_hp.pdf; and with no valid negative mammography results as defined by CEWG).
Risk level of hypertension | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The hypertension risk level will be defined as low-risk with SBP≤120 mmHg, and DBP ≤ 80 mmHg; medium-risk with SBP 120-139 mmHg, and/or DBP 80-89 mmHg; high risk with Systolic Blood Pressure (SBP) ≥ 140 mmHg, and/or Diastolic Blood Pressure (SBP) ≥ 90 mmHg. The classification is based on seated clinic blood pressure. If SBP and DBP fall into different categories, the higher category should be used to classify blood pressure risk level. Three seated clinic BP measurements will be recorded, 1-2 min apart, and additional measurements only if the first two readings differ by &amp;amp;amp;amp;amp;amp;amp;amp;amp;gt;10 mmHg. BP is recorded as the average of the last two BP readings.
Risk level of cervical cancer | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The cervical cancer risk level will be assessed using the risk assessment questionnaire covering the HK CEWG risk factors (as described in https://www.chp.gov.hk/files/pdf/cervical_cancer_professional_hp.pdf). Risk levels are categorized as low (women never had any sexual experience, and are not vulnerable to HPV infection and with no risk factors; or those who have valid negative screening results as defined by CEWG), medium (women never had any sexual experience, and are not vulnerable to HPV infection, and with risk factors of tobacco use/long term use of oral contraceptives for non-medical indication), high ( women had sexual experience (e.g., non-penetrative, penetrative, vaginal, oral, anal sex), and/or are vulnerable to Human Papillomavirus (HPV) infection by meeting the risk factors (e.g. immunocompromised individuals, recipients of organ transplant, with STIs co-infection), and have no valid negative screening results as defined by CEWG).
Risk level of colorectal cancer | 1- , 3-, 6-, 7-, and 12-month after baseline.
  The colorectal cancer risk level will be assessed using the risk assessment questionnaires covers the risk factors (as described in https://www.chp.gov.hk/files/pdf/cewg_crc_professional_hp.pdf and https://www.colonscreen.gov.hk). Risk levels are categorized as low (women aged below 50, and without disease-related risk factors and lifestyle modifiable risk factors; or anyone has valid negative cancer screening result), medium (women aged below 50, and without disease-related risk factors, and with any one of the modifiable risk factors), high (women aged ≥ 50 years old, or anyone meets HK CEWG increased risk definitions, or anyone has symptoms of colorectal cancer/ history of colorectal cancer/ history of chronic inflammation of the bowel (e.g. ulcerative colitis)/ diagnosis of hereditary bowel syndromes/ family history of first-degree relative having hereditary bowel syndromes/ history of colorectal polyps; and have no valid negative cancer screening results).

CONTACTS AND LOCATIONS:
Overall Officials: Siu Chee Chan, Professor, Principal Investigator — The University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Aberdeen Kaifong Welfare Association, Hong Kong
  - Haven of Hope Christian Service, Hong Kong
  - Hong Kong Sheng Kung Hui Welfare Council, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data collected during the trial will be shared at 2 years after article publication with no end date.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Nasreen SZA: Management of Menopause: Jaypee Brothers Medical Publishers; 2021.
- [Background] Saitz R, Alford DP, Bernstein J, Cheng DM, Samet J, Palfai T. Screening and brief intervention for unhealthy drug use in primary care settings: randomized clinical trials are needed. J Addict Med. 2010 Sep;4(3):123-30. doi: 10.1097/ADM.0b013e3181db6b67. PMID 20936079
- [Background] Slev VN, Molenkamp CM, Eeltink CM, Roeline W Pasman H, Verdonck-de Leeuw IM, Francke AL, van Uden-Kraan CF. A nurse-led self-management support intervention for patients and informal caregivers facing incurable cancer: A feasibility study from the perspective of nurses. Eur J Oncol Nurs. 2020 Apr;45:101716. doi: 10.1016/j.ejon.2019.101716. Epub 2020 Jan 20. PMID 32023503
- [Background] Kolac N, Yildiz A. The effect of health belief model-based short interviews in women in the postmenopausal period on the prevention of osteoporosis: A randomized controlled trial. Int J Nurs Pract. 2023 Feb;29(1):e13121. doi: 10.1111/ijn.13121. Epub 2022 Dec 16. PMID 36524466
- [Background] Wang MP, Luk TT, Wu Y, Li WH, Cheung DY, Kwong AC, Lai V, Chan SS, Lam TH. Chat-based instant messaging support integrated with brief interventions for smoking cessation: a community-based, pragmatic, cluster-randomised controlled trial. Lancet Digit Health. 2019 Aug;1(4):e183-e192. doi: 10.1016/S2589-7500(19)30082-2. Epub 2019 Jul 31. PMID 33323188
- [Background] Li C, Liu Y, Xue D, Chan CWH. Effects of nurse-led interventions on early detection of cancer: A systematic review and meta-analysis. Int J Nurs Stud. 2020 Oct;110:103684. doi: 10.1016/j.ijnurstu.2020.103684. Epub 2020 Jun 12. PMID 32702568
- [Background] Chłoń-Domińczak A, Kotowska IE, Kurkiewicz J, Abramowska-Kmon A, Stonawski M: Population ageing in Europe: facts, implications and policies. Brussels: European Commission 2014
- [Background] United Nations. World Population Ageing 2017 Highlights (ST/ESA/SER.A/397). Population Division World Population Ageing. 2017.